CLINICAL TRIAL: NCT05313828
Title: Effect of Various Treatment Modalities on Dendritic Vial Ulcer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Mahmoud,MD, principal investigator, Sohag University
Other Study IDs: soh-med-22-02-28
Record Dates: First submitted 2022-03-26; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer | interventions — Acyclovir; Tobramycin; Fluorometholone; Hyaluronic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 1': patients with viral ulcers will receive antiviral medication with antibiotics
  Interventions: Drug: Acyclovir; Drug: Tobramycin
- group 2: patients with viral ulcers will receive antiviral medication, tear substitutes with antibiotics
  Interventions: Drug: Acyclovir; Drug: Tobramycin; Drug: Sodium Hyaluronate
- group 3: patients with viral ulcers will receive antiviral medication, weak steroids(at the same time) with antibiotics
  Interventions: Drug: Acyclovir; Drug: Tobramycin; Drug: Fluorometholone
- group 4: patients with viral ulcers will receive antiviral medication with antibiotics followed by weak steroid after epithelial healing
  Interventions: Drug: Acyclovir; Drug: Tobramycin; Drug: Fluorometholone

INTERVENTIONS:
Drug: Acyclovir — acyclovir 4 times /day
Drug: Tobramycin — tobramycin 4 times /day
Drug: Fluorometholone — Fluorometholone 4 times/ day
  Groups: group 3; group 4
Drug: Sodium Hyaluronate — Sodium Hyaluronate 4 times/day
  Groups: group 2

SUMMARY:
Eye infection is a prevalent problem in primary care and remains a crucial healthcare concern. According to the American Academy of Ophthalmology (AAO), herpes simplex virus (HSV) keratitis (HSK) is the leading cause of infectious blindness worldwide . HSK is defined as a corneal inflammatory condition caused by the HSV infection . The global incidence of herpetic keratitis is estimated at 1.5 million per year, resulting in 40,000 new cases of severe visual impairment associated with corneal scarring and opacification . HSV type I (HSV-1) is by far the most predominant causative pathogen of eye infections]. HSV-1 is also known for causing orolabial herpes, HSV folliculitis, herpes gladiatorum, herpetic whitlow, and eczema herpeticum . HSV can be transferred to the eye by touching an active lesion and then the eye. The National Health and Nutrition Evaluation revealed a seroprevalence of HSV-1 in 53.9% of 14-49 year olds, and 90% of adults 50 years or older , indicating that the majority of the population has been exposed to this virus thus are at risk of developing HSK.

In this study we evaluate the efficacy of different treatment modalities on viral keratitis HSK.

ELIGIBILITY:
Inclusion Criteria:

patients with epithelial viral ulcers

-

Exclusion Criteria:

* patients with stromal keratitis patients with corneal opacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from epithelial viral keratitis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-06-28 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
healing of the epithelium | 10 days follow up
  the epithelial healing assessed with flourescin stain and measured by slit lamp scale in millimetres and compared with pre treatment epithelial defect

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code